CLINICAL TRIAL: NCT00133172
Title: Evaluation of the Long-term Safety and Efficacy of a Tacrolimus-based 5-day Steroid Rapid Withdrawal Immunoprophylactic Regimen in de Novo Renal Transplantation
Brief Title: Effect of Rapid Steroid Withdrawal on Subclinical Markers of Rejection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Varience of supply chain from that required by protocol
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FKC-011
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Kidney Transplantation
Keywords: Treatment Efficacy; Treatment Effectiveness; Anti-rejection therapy; Immunosuppression; Antirejection; Renal Transplantation; Transplantation, Renal; Transplantation, Kidney; Grafting, Kidney
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Steroid rapid 5-day withdrawal
  Interventions: Drug: Tacrolimus; Drug: mycophenolate mofetil; Drug: Prednisone
- 2 (Active Comparator): Standard steroid maintenance
  Interventions: Drug: Tacrolimus; Drug: mycophenolate mofetil; Drug: Prednisone

INTERVENTIONS:
Drug: Tacrolimus — IV
  Other Names: Prograf; FK506
Drug: mycophenolate mofetil — IV
  Other Names: Cellcept
Drug: Prednisone — IV

SUMMARY:
The purpose of this study is to compare the safety and efficacy of a tacrolimus-based 5-day steroid rapid withdrawal immunoprophylactic regimen in de novo renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally acceptable guardian has signed and dated a Research Ethics Board (REB)-approved informed consent form and is willing and able to follow study procedures.
* Subject is the recipient of a first or second cadaveric or living donor mismatched (at least one mismatch) renal transplant.
* Subject is 18 years of age or over at the time of transplant.
* If female and of child-bearing potential, subject has a negative pregnancy test and utilizes adequate contraceptive methods

Exclusion Criteria:

* Recipients of a kidney from a donor 60 years of age or older
* Recipients of donation after cardiac death (DCD) donors
* Recipients of a combined transplant (e.g. kidney-pancreas, -lung, -heart)
* Subjects with a second renal allograft who had their original graft for < 2 years, unless the initial graft was lost in the early (1 year or less) post transplant course due to a technical or surgical failure
* Subjects with a current/latest pre-transplant panel of reactive antibodies (PRA) >20
* Subjects with hepatitis B & C, HIV or cancer (excluding successfully excised squamous or basal cell carcinoma)
* Subjects receiving an allograft with cold ischemia time 24 hours or greater
* Subjects who have received an investigational drug within three months prior to randomization
* Subjects who are breastfeeding
* Subjects with known hypersensitivity to tacrolimus, mycophenolate mofetil, methylprednisolone, basiliximab, prednisone, or any related drugs or their excipients
* Subjects with significant disease (e.g. uncontrolled infection) or disability (e.g. cognitive deficit) that prevents understanding of or adherence to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Combined incidence of biopsy proven subclinical rejection (BPSCR) and biopsy proven clinical acute rejection (BPCAR) | 3 months post transplant

SECONDARY OUTCOMES:
Biopsy proven chronic allograft nephropathy(CAN) | 2 years post transplant
Patient and graft survival rates | End of study (5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Canada, Inc.
Locations (10):
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan